CLINICAL TRIAL: NCT03071640
Title: Improving Quality of Life and Function for Older Cancer Patients Receiving Radiotherapy. Part IC: A Prospective Observational Study
Brief Title: Improving Quality of Life and Function for Older Cancer Patients Receiving Radiotherapy
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Norwegian University of Science and Technology (Other); St. Olavs Hospital (Other); Oslo University Hospital (Other); Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: 150356
Record Dates: First submitted 2017-02-16; First posted 2017-03-07 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2019-10

CONDITIONS: Elderly; Cancer; Radiotherapy Side Effect
Keywords: old; elderly; radiotherapy; geriatric assessment
MeSH Terms: conditions — Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a first part of a larger project aiming at improving the following outcomes in older cancer patients receiving external beam radiation therapy (EBRT): quality of life, functioning and need for professional help (dependency). To achieve this, the investigators will develop and test a geriatric assessment (GA) with management (GAM) intervention targeting patients at risk of negative outcomes as defined. The problems and needs that older patients experience before, during and after EBRT are poorly described. Furthermore, although GA is the recommended approach to assess older cancer patients' vulnerability, very few studies have investigated its benefit and feasibility in a radiotherapy setting and there is no universal recipe for how an efficient GAM intervention should be applied in this setting. Before defining and testing an intervention, the investigators will therefore conduct an observational study addressing older patients >= 65 years referred for either palliative or curative EBRT. The main objectives are to identify patients at risk for negative outcomes, and to test the feasibility of GA in the community service and at a radiotherapy department.

DETAILED DESCRIPTION:
GA includes a systematic assessment of area where older people often have problems, i.e. assessment of comorbidity, medication, functional status and physical functioning, cognitive function, nutritional status, and depression. In this observational study, the assessment will be performed using well-established instruments and tests before start and after completion of radiotherapy. The patient will be followed-up by repeated assessments at week 2, 8 and 16 post treatment. Quality of life (QoL) questionnaires will be filled in by self-report at the same points in time. Follow-up data will also include information on the patients' use of health services (home-, nursing home and hospital care). Additionally available diagnostic CT scans will also be used for analyses of nutritional status and body composition. Eligible patients will be included at the Radiotherapy Unit, Innlandet Hospital Trust after having given written informed consent. A project nurse (cancer nurse) will perform the assessments at the Radiotherapy Unit, whereas follow-up assessments will be performed by community cancer nurses. All municipalities in the hospital catchment area are invited to participate in the study. The study will be conducted in co-operation with several national and international partners, including partners from the local municipalities

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 65 years of age
* histologically confirmed cancer diagnoses
* referred for palliative or curative EBRT
* living in the hospital catchment area, able to understand and fill in self-report questionnaires
* fluent in Norwegian (orally and in writing), provide written, informed consent

Exclusion Criteria:

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients >= 65 years of age referred for palliative or curative EBRT at the Radiotherapy Unit, Innlandet Hospital Trust
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2020-07-19 (Actual)

PRIMARY OUTCOMES:
physical function | within 16 weeks after completion of EBRT
  as measured by the EORTC QLQ-C30
global quality of life | within 16 weeks after completion of EBRT
  as measured by the EORTC QLQ-C30

SECONDARY OUTCOMES:
Dependency | within 16 weeks after completion of EBRT
  As measured by the Nottingham Extended Activities of Daily Living
Use of inpatient services | within 16 weeks after completion of EBRT
  inpatient days, hospital and nursing homes

OTHER OUTCOMES:
Feasibility of GA | within 16 weeks after completion of EBRT
  Registered by questionnaires to participating cancer nurses
Edmonton Frail Scale | baseline and within 16 weeks after completion of EBRT
  the precision of Edmonton Frail Scale in detecting frailty will be tested as compared to the more comprehensive GA

CONTACTS AND LOCATIONS:
Overall Officials: Marit Jordhøy, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- The Radiotherapy Unit, Innlandet Hospital Trust, Gjøvik, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eriksen GF, Benth JS, Gronberg BH, Rostoft S, Kirkhus L, Kirkevold O, Oldervoll LM, Bye A, Hjelstuen A, Slaaen M. Geriatric impairments are associated with reduced quality of life and physical function in older patients with cancer receiving radiotherapy - A prospective observational study. J Geriatr Oncol. 2023 Jan;14(1):101379. doi: 10.1016/j.jgo.2022.09.008. Epub 2022 Sep 27. PMID 36180379
- [Derived] Eriksen GF, Saltyte Benth J, Gronberg BH, Rostoft S, Kirkevold O, Bergh S, Hjelstuen A, Rolfson D, Slaaen M. Cognitive Trajectories in Older Patients with Cancer Undergoing Radiotherapy-A Prospective Observational Study. Curr Oncol. 2022 Jul 21;29(7):5164-5178. doi: 10.3390/curroncol29070409. PMID 35877269
- [Derived] Eriksen GF, Saltyte Benth J, Gronberg BH, Rostoft S, Kirkhus L, Kirkevold O, Hjelstuen A, Slaaen M. Geriatric impairments are prevalent and predictive of survival in older patients with cancer receiving radiotherapy: a prospective observational study. Acta Oncol. 2022 Apr;61(4):393-402. doi: 10.1080/0284186X.2021.2009561. Epub 2021 Dec 7. PMID 34874228

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT03071640/Prot_SAP_000.pdf